CLINICAL TRIAL: NCT04183296
Title: The Effect of Total Intravenous Anesthesia and Volatile Anesthesia on Shedding of the Endothelial Glycocalyx in Patients Undergoing Laparoscopic or Robotic Assisted Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 4-2019-0924
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Gastrostomy
Keywords: Laparoscopic assisted gastrectomy; Robotic assisted gastrectomy
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: A Randomized Trial
Masking Description: triple (Participant, Care Provider, investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA(Total Intravenous Anesthesia and Volatile Anesthesia ) (Experimental): In the TIVA group, anesthesia was induced with TCI of propofol (Ce of 4.0-4.5 μg/ml) and remifentanil (Ce of 4.0 ng/ml). Anesthesia was maintained with TCI of propofol and remifentanil. Anesthesia depth was adjusted to maintain a PSI of 25-50.
  Interventions: Drug: propofol
- Inhalation (Active Comparator): Arm Description: In the volatile group, anesthesia was induced with an intravenous bolus of propofol 1.5-2 mg/kg and TCI of remifentanil (effect-site concentration [Ce] of 4.0 ng/ml). Anesthesia was maintained with sevoflurane (0.8-1 age-adjusted minimum alveolar concentration) and TCI of remifentanil
  Interventions: Drug: sevoflurane

INTERVENTIONS:
Drug: propofol — Anesthesia was induced with TCI of propofol (Ce of 4.0-4.5 μg/ml) and remifentanil (Ce of 4.0 ng/ml). Anesthesia was maintained with TCI of propofol and remifentanil. Anesthesia depth was adjusted to maintain a PSI of 25-50.
  Other Names: TIVA group
  Arms: TIVA(Total Intravenous Anesthesia and Volatile Anesthesia )
Drug: sevoflurane — Anesthesia was induced with an intravenous bolus of propofol 1.5-2 mg/kg and TCI of remifentanil (effect-site concentration [Ce] of 4.0 ng/ml). Anesthesia was maintained with sevoflurane (0.8-1 age-adjusted minimum alveolar concentration) and TCI of remifentanil
  Other Names: volatile group
  Arms: Inhalation

SUMMARY:
The aim of this study was to investigate the effects of total intravenous and inhalation anesthesia on the damage of endothelial glucocorticoids by comparing the concentration of syndecan-1 before and after laparoscopic or robotic assisted gastrectomy.

DETAILED DESCRIPTION:
A commercial TIVA(Total Intravenous Anesthesia and Volatile Anesthesia ) pump was used for target-controlled infusion (TCI) of remifentanil and propofol. In the volatile group, anesthesia was induced with an intravenous bolus of propofol 1.5-2 mg/kg and TCI of remifentanil (effect-site concentration [Ce] of 4.0 ng/ml). In the TIVA group, anesthesia was induced with TCI of propofol (Ce of 4.0-4.5 μg/ml) and remifentanil (Ce of 4.0 ng/ml). In the volatile group, anesthesia was maintained with sevoflurane (0.8-1 age-adjusted minimum alveolar concentration [MAC]) and TCI of remifentanil, while in the TIVA group, anesthesia was maintained with TCI of propofol and remifentanil. Anesthesia depth was adjusted to maintain a PSI(Patient State Index) of 25-50. Endotracheal intubation was performed after administration of intravenous rocuronium 1.2 mg/kg and neuromuscular blockade depth was maintained to a target of train-of-four of 0-2 with infusion of rocuronium during pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients over 20 years old with ASA class I-III
2. Scheduled laparoscopic or robotic assisted laparoscopic gastrectomy

Exclusion Criteria:

1. emergency surgery
2. patients unable to make their own decisions, illiterate, foreigners
3. Allergy / hypersensitivity to sevoflurane or propofol 4, Current or past history or thrombosis / thromboembolism

5. patients who are taking oral contraceptives 6. Patients with renal insufficiency (eGFR 60 ml / min / 1.73 m 2 or less) 7. Patients receiving anticoagulants 8. pregnant and lactating women 9. Patients with history of psychiatric disease or neurological disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-11-28 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Changes in blood concentration of syndecan-1 | after anesthesia induction <before surgery(base concentration)>
  Blood levels of syndecan-1 are assessed at 10 minutes after anesthesia induction.
Changes in blood concentration of syndecan-1 | at the end of surgery
  Blood levels of syndecan-1 are assessed at the end of surgery.
Changes in blood concentration of syndecan-1 | 1 day after surgery
  Blood levels of syndecan-1 are assessed 1 day after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim NY, Kim KJ, Lee KY, Shin HJ, Cho J, Nam DJ, Kim SY. Effect of volatile and total intravenous anesthesia on syndecan-1 shedding after minimally invasive gastrectomy: a randomized trial. Sci Rep. 2021 Jan 15;11(1):1511. doi: 10.1038/s41598-021-81012-1. PMID 33452350